CLINICAL TRIAL: NCT02494219
Title: Comparison of Immunochromatographic Test for Rapid Detection of Group A Streptococcal Antigen With Culture in Pediatric Patients
Brief Title: Pharyngitis,Group A Streptococcal Infection,Rapid Streptococcal Test,Throat Swab Culture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HamadMC
Record Dates: First submitted 2015-06-18; First posted 2015-07-10 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-06

CONDITIONS: Pharyngitis
Keywords: Group A streptococcal pharyngitis; Rapid streptococcal test; Throat swab culture
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rapid Immunochromatographic Streptococcal test (Experimental): Throat swabbing by two port germ Amines agar (copan) swabs,the swabs were randomly labeled as swab A and swab B.Swab A was processed for rapid streptococcal test and swab B was processed for culture in Colombia blood agar.All patients were followed up after 48-72 hours with the final culture results that ultimately determined the need to continue or discontinue treatment.
  Interventions: Procedure: Rapid Immunochromatographic streptococcal test

INTERVENTIONS:
Procedure: Rapid Immunochromatographic streptococcal test — Throat swab obtained for rapid strep test in addition to throat culture,in order to check the accuracy of Rapid Immunochromatographic streptococcal test in detection of streptococcal pharyngitis

SUMMARY:
Comparison of Immunochromatographic Test for rapid detection of group A streptococcal antigen with culture in Pediatric patients.

DETAILED DESCRIPTION:
Throat swabbing by two port germ Amines agar (copan) swabs,then the swabs were randomly labeled as swab A and swab B.Swab A was processed for rapid streptococcal test and swab B was processed for culture in Colombia blood agar.All patients were followed up after 48-72 hours with the final culture results that ultimately determined the need to continue or discontinue treatment.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting with the possible diagnosis of Bacterial pharyngitis,between 1-14 years of age.

Exclusion Criteria:

* Patients who received antibiotics within two weeks from presentation

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 906 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The ratio of true negative rapid immunochromatographic strep test when compared throat culture | upto 48 hours

SECONDARY OUTCOMES:
The ratio of true positive rapid immunochromatographic strep test when compared to throat culture | upto 48hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad medical corporation, Doha, Qatar